CLINICAL TRIAL: NCT03132441
Title: A Prospective Trial to Evaluate the Utility of Focused Frailty Interventions on Patients Undergoing Evaluation for Left Ventricular Assist Device (LVAD) Placement
Brief Title: Cardiac Rehab for Advanced Heart Failure-LVAD Candidates
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Major changes to study that were better suited to creating a whole new study
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sudhir Kushwaha, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-000210
Record Dates: First submitted 2017-04-25; First posted 2017-04-27 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Heart Failure
Keywords: advanced heart failure; NYHA Class III-IV; frailty; cardiac rehabilitation
MeSH Terms: conditions — Heart Failure; Frailty | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Single arm pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac Rehabilitation (Experimental): Strength Training for Frailty:
  All patients enrolled will be enrolled in 6 weeks of cardiac rehabilitation for the pilot study.
  Interventions: Other: Strength Training for Frailty

INTERVENTIONS:
Other: Strength Training for Frailty — Cardiac Rehabilitation, abbreviated course

SUMMARY:
This study is a pilot study evaluating the feasibility and early efficacy of cardiac rehabilitation to improve frailty and symptoms in patients with advanced heart failure (NYHA class III-IV), who are being considered for LVAD therapy.

DETAILED DESCRIPTION:
Frailty in patients with advanced heart failure is not thoroughly described, but in those studies that assessed frailty, it was a common phenomenon. Furthermore, some data suggest an association between pre-LVAD implant frailty and post-implant complications and survival. Interventions for frailty have been utilized in various populations, including the elderly frail and the frail from cardiovascular causes. These interventions target physical strengthening and endurance and have been shown on occasion to improve functional outcomes. The current study, a pilot study, seeks to assess frailty in a prospective cohort of patients being evaluated in Heart Failure Clinic for consideration of LVAD implantation due to NYHA class III-IV dyspnea and enroll these patients in a six-week focused cardiac rehabilitation protocol aimed at improving frailty and functional independence. The primary endpoint of the study is improvement in frailty markers at the end (gait speed, handgrip strength), and secondary endpoints include improvement in the indices of quality of life and symptomatology via validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for a Left Ventricular Assist Device (LVAD)
* Advanced Heart Failure as determined by New York Heart Association classification III or IV

Exclusion Criteria:

* Unable to perform physical activities required by protocol due to anatomic or musculoskeletal comorbidities
* Physical activity is contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04 (Estimated); Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Change in frailty marker handgrip strength | Baseline, 6 weeks
  Frailty is assessed by the strength of a participant's handgrip, measured using a commercial device.
Change in frailty marker gait speed | Baseline, 6 weeks
  Frailty is assessed by the strength of a participant's gait speed, measured using a commercial device.

SECONDARY OUTCOMES:
Change in New York Heart Association (NYHA) classification | Baseline, 6 weeks
  New York Heart Association (NYHA) Classification Scale Early-Stage Heart Failure
  * NYHA Class I No symptoms at any level of exertion and no limitation in ordinary physical activity.
  * NYHA Class II Mild symptoms and slight limitation during regular activity. Comfortable at rest.
  Advanced-Stage Heart Failure
  * NYHA Class III Noticeable limitation due to symptoms, even during minimal activity. Comfortable only at rest.
  * NYHA Class IV Severe limitations. Experience symptoms even while at rest (sitting in a recliner or watching TV).
Change in Minnesota Living with Heart Failure (MLHF) score | Baseline, 6 weeks
  A participant's quality of life assessed by Minnesota Living with Heart Failure (MLHF) questionnaire score.
Change in KCCQ score | Baseline, 6 weeks
  A participant's quality of life assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ) questionnaire score.

CONTACTS AND LOCATIONS:
Overall Officials: Sudhir S Kushwaha, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic-Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh M, Stewart R, White H. Importance of frailty in patients with cardiovascular disease. Eur Heart J. 2014 Jul;35(26):1726-31. doi: 10.1093/eurheartj/ehu197. Epub 2014 May 26. PMID 24864078
- [Background] Dunlay SM, Park SJ, Joyce LD, Daly RC, Stulak JM, McNallan SM, Roger VL, Kushwaha SS. Frailty and outcomes after implantation of left ventricular assist device as destination therapy. J Heart Lung Transplant. 2014 Apr;33(4):359-65. doi: 10.1016/j.healun.2013.12.014. Epub 2013 Dec 27. PMID 24486165
- [Background] Thalji NM, Suri RM, Greason KL, Schaff HV. Risk assessment methods for cardiac surgery and intervention. Nat Rev Cardiol. 2014 Dec;11(12):704-14. doi: 10.1038/nrcardio.2014.136. Epub 2014 Sep 23. PMID 25245832
- [Background] Flint KM, Matlock DD, Lindenfeld J, Allen LA. Frailty and the selection of patients for destination therapy left ventricular assist device. Circ Heart Fail. 2012 Mar 1;5(2):286-93. doi: 10.1161/CIRCHEARTFAILURE.111.963215. No abstract available. PMID 22438521
- [Background] Chung CJ, Wu C, Jones M, Kato TS, Dam TT, Givens RC, Templeton DL, Maurer MS, Naka Y, Takayama H, Mancini DM, Schulze PC. Reduced handgrip strength as a marker of frailty predicts clinical outcomes in patients with heart failure undergoing ventricular assist device placement. J Card Fail. 2014 May;20(5):310-5. doi: 10.1016/j.cardfail.2014.02.008. Epub 2014 Feb 22. PMID 24569037
- [Background] Molino-Lova R, Pasquini G, Vannetti F, Paperini A, Forconi T, Polcaro P, Zipoli R, Cecchi F, Macchi C. Effects of a structured physical activity intervention on measures of physical performance in frail elderly patients after cardiac rehabilitation: a pilot study with 1-year follow-up. Intern Emerg Med. 2013 Oct;8(7):581-9. doi: 10.1007/s11739-011-0654-z. Epub 2011 Jul 9. PMID 21744061